CLINICAL TRIAL: NCT01487798
Title: A Double-blind, Randomised, Crossover Study to Investigate the Difference in Frequency of Episodes of Hypoglycaemia During Treatment With Biphasic Insulin Aspart 30 Compared to Biphasic Human Insulin 30 in Patients With Well-controlled Type 2 Diabetes
Brief Title: Frequency of Episodes of Hypoglycaemia During Treatment With Biphasic Insulin Aspart 30 in Type 2 Diabetes
Acronym: REACH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1466
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — biphasic human insulin 30; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: biphasic human insulin 30; Drug: biphasic insulin aspart 30
- Treatment period 2 (Active Comparator)
  Interventions: Drug: biphasic human insulin 30; Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic human insulin 30 — Administrated s.c. (subcutaneously, under the skin) for 16 weeks in treatment period 1 followed by 16 weeks in treatment period 2
Drug: biphasic insulin aspart 30 — Administrated s.c. (subcutaneously, under the skin) for 16 weeks in treatment period 1 followed by 16 weeks in treatment period 2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the difference in frequency of episodes of hypoglycaemia during treatment with biphasic insulin aspart 30 compared to biphasic human insulin 30 in subjects with well controlled type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treated with insulin 1-3 injections daily for at least 6 months
* Body Mass Index (BMI) below 40 kg/m^2
* HbA1c (glycosylated haemoglobin A1c) below 9.5% at screening

Exclusion Criteria:

* Total insulin dosage more than 1.8 IU/kg
* Impaired hepatic or renal function or significant cardiac problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2002-06; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Frequency of hypoglycaemic episodes

SECONDARY OUTCOMES:
Frequency of reported severe hypoglycaemic episodes
Overall frequency of nocturnal hypoglycaemia
HbA1c (glycosylated haemoglobin A1c)
Diabetes Treatment Satisfaction Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (16):
- United Kingdom (16):
  - Novo Nordisk Investigational Site, Bolton
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, Derby
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Exeter
  - Novo Nordisk Investigational Site, Galway
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Newcastle
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Upton
  - Novo Nordisk Investigational Site, Wirral, Merseyside
  - Novo Nordisk Investigational Site, York

REFERENCES:
- [Result] McNally PG, Dean JD, Morris AD, Wilkinson PD, Compion G, Heller SR. Using continuous glucose monitoring to measure the frequency of low glucose values when using biphasic insulin aspart 30 compared with biphasic human insulin 30: a double-blind crossover study in individuals with type 2 diabetes. Diabetes Care. 2007 May;30(5):1044-8. doi: 10.2337/dc06-1328. Epub 2007 Feb 2. PMID 17277042
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com